CLINICAL TRIAL: NCT04473950
Title: The Effect of Chronic Pain on Delay Discounting in Methadone Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The COVID-19 Pandemic prevented us from meeting target goals.
Sponsor: University of California, San Francisco (Other)
Collaborators: Johns Hopkins University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Z-1902; R21DA047520 (NIH)
Record Dates: First submitted 2020-06-12; First posted 2020-07-16 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Opioid-use Disorder; Chronic Pain Syndrome
Keywords: delay discounting; pain catastrophizing; impulsivity
MeSH Terms: conditions — Opioid-Related Disorders; Impulsive Behavior | interventions — Naloxone

STUDY DESIGN:
Intervention Model Description: This proposal is a randomized double-blind placebo controlled Phase 1 clinical trial / human laboratory study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, investigator, medical personnel administering study drug, and outcomes assessor will be blinded to drug being administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pain Group (Experimental): Patients with chronic pain who are maintained on methadone for opioid use disorder
  Interventions: Drug: Naloxone Hydrochloride; Drug: Placebo
- No Pain Group (Placebo Comparator): Patients who are maintained on methadone for opioid use disorder but who do not have chronic pain.
  Interventions: Drug: Naloxone Hydrochloride; Drug: Placebo

INTERVENTIONS:
Drug: Naloxone Hydrochloride — An intramuscular (IM) injection of naloxone will be given.
  Other Names: Narcan
Drug: Placebo — An IM injection of 0.9% normal saline will be given.

SUMMARY:
The epidemic of opioid overdose deaths continues to rise, killing more persons in 2017 than HIV/AIDS at the height of that epidemic. Medication assisted treatment, including methadone and buprenorphine, is the standard of care for the treatment of opioid use disorder (OUD). However, chronic pain can reduce treatment efficacy during medication assisted treatment and is associated with illicit substance relapse, dropout, and subsequent overdose. Mechanisms by which chronic pain may influence the impulsive decision making (e.g., drug relapse) in persons with OUD have not been well characterized. A better understanding is needed of decision-making in this population. Two factors that can influence decisions to use drugs are impulsivity and acute opioid withdrawal. This proposal will test how chronic pain is associated with increases in impulsive decision making in OUD, whether impulsive decision making is greater when undergoing opioid withdrawal, and how catastrophizing may modify the association between withdrawal and impulsive decision making in patients with chronic pain and OUD. An ideal population for this developmental research project are methadone maintained patients, who show high treatment attendance rates and will therefore assure study efficiency and reliable completion.

DETAILED DESCRIPTION:
This is an outpatient Phase 1 clinical trial investigating the effect of naloxone precipitated withdrawal on delay discounting. Eligible participants will undergo two experimental sessions presented in random order. One session will involve the measurement of delay discounting 30 minutes after double-blind intramuscular (IM) administration of placebo (normal saline) and the other will have the exact same procedures performed after double-blind IM administration of naloxone (0.1 mg). Injections will occur 2 hours after methadone dosing (peak levels). Study sessions will last 2 hours and involve pain and opioid withdrawal measures assessed at baseline and 15 minute intervals after injections. The participant should be back to baseline and free of withdrawal by the end of the study session. Sessions will occur at least 48 hours apart.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged 18-65
* Stable methadone dose (at least 21 days) verified by contacting participant's opioid treatment program
* Understand and speak English
* Urine toxicology screen negative for drugs of abuse and positive for methadone
* Participants must be without signs of intoxication as evidenced by ability to receive full dose of methadone prior to research activities.
* Presence of chronic pain (>3 months) for the Pain group and absence of pain for the No Pain group.

Exclusion Criteria:

* Unstable psychiatric illness as assessed by the Mini International Neuropsychiatric Interview (e.g. active suicidal ideation, psychosis)
* Unstable medical illness as assessed by the study's independent medical monitor (e.g. uncontrolled hypertension, recent myocardial infarction, recent stroke, unstable angina) that may be affected by precipitated withdrawal
* Prescription opioid use besides methadone
* Acute pain process unrelated to chronic pain
* Women who are pregnant or lactating
* Known allergy to naloxone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D. Andrew Tompkins, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to the public through presentation at scientific meetings and research publications in peer-reviewed journals. I have routinely kept an open policy to share data with the scientific and medical community upon request, and this policy will be continued with the present project.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available after publication of the main study results.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We began study recruitment in January 2020 (Q2) after IRB approval was received. The first study participant screening session was on January 21, 2020. UCSF halted all non-essential clinical research in March 2020 and we were unable to conduct research activities on a full 5 day a week schedule until one year later, with some periods during winter surges when we had to again shut down all research activities.
Period: Overall Study
Arm/Group | Pain Group | No Pain Group
Started | 6 | 4
Naloxone | 6 | 4
Placebo | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pain Group | No Pain Group | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.83 (10.98) | 38.25 (7.46) | 47.6 (12.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Delay Discounting of Money Rate (k)
Description: Delay discounting is the relative preference for smaller sooner over larger later rewards, an aspect of impulsivity. Most individuals would prefer an immediate $100 over $100 delayed by 1 year. However, when faced with the choice between receiving $95 now versus $100 in 1 year, preferences for the delayed reward may increase. By assessing such choices across multiple delays, delay discounting quantifies the devaluation of rewards over time, which allows for an index of overall discounting rate (k). Delay Discounting of money rate has no units and values can go from 0-infinity. A larger discount rate indicates that a future reward is devalued more, and is associated with more impulsive behavior.
Time Frame: k will be calculated from the same series of discounting questions that will be asked once each session at approximately 30 minutes after study medication administration.
Measure: Mean (Standard Deviation); unit: k-value
Arm/Group | Pain Group | No Pain Group
Number analyzed (Participants) | 6 | 4
k-value
  Naloxone Session | -1.65 (1.17) | -2.16 (0.92)
  Placebo Session | -1.91 (0.56) | -2.11 (1.11)

2. Secondary Outcome: Study Session Peak Pain Visual Analog Scale (VAS)
Description: Current pain level rated on 0-100 VAS. This is the validated pain scale typically used by clinicians in an outpatient or inpatient clinical visit to represent current level of pain. Higher ratings indicate worse pain severity.
Time Frame: Peak Pain VAS will be the highest rating during each 2 hour study session.
Population: There was missing data for one participant with chronic pain in the placebo session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Group | No Pain Group
Number analyzed (Participants) | 6 | 4
score on a scale
  Placebo: number analyzed (Participants) | 5 | 4
  Placebo | 25.2 (22.9) | 0 (0)
  Naloxone | 28.2 (25.4) | 0.25 (0.5)

3. Secondary Outcome: Peak Clinical Opiate Withdrawal Scale (COWS) Rating
Description: The COWS is an 11-item validated clinician administered scale that quantifies level of opioid withdrawal. The range of scores is 0-48, with higher scores indicating greater withdrawal severity. The peak COWS rating will be the highest measurement in the session after study drug administration.
Time Frame: Peak COWS rating will be the highest rating during each 2 hour study session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Group | No Pain Group
Number analyzed (Participants) | 6 | 4
score on a scale
  Placebo | 1.8 (0.98) | 2.75 (0.5)
  Naloxone | 2.5 (2.6) | 3 (2.4)

4. Secondary Outcome: Peak Subjective Opiate Withdrawal Scale (SOWS) Rating
Description: The SOWS is a 16 item validated self-administered scale for grading opioid withdrawal symptoms. The range of scores is 0-64, with higher scores indicating greater withdrawal severity. The peak SOWS rating will be the highest measurement in the session after study drug administration.
Time Frame: Peak SOWS rating will be the highest rating during each 2 hour study session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Group | No Pain Group
Number analyzed (Participants) | 6 | 4
score on a scale
  Placebo | 3.2 (2.6) | 2.8 (2.1)
  Naloxone | 2.7 (2.9) | 3.8 (2.1)

5. Secondary Outcome: Peak Increase From Baseline Pupil Diameter
Description: Pupil diameter (mm) will be measured via digital pupillometer in standard room lighting at baseline and then throughout the study session after study drug administration. The peak increase from baseline value will be the largest increase from baseline pupil diameter measured after study drug administration.
Time Frame: Peak increase from baseline pupil diameter will be the largest increase from baseline pupil diameter measured during each 2 hour study session.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Pain Group | No Pain Group
Number analyzed (Participants) | 6 | 4
millimeters
  Placebo | 0.06 (0.08) | 0.03 (0.07)
  Naloxone | 0.31 (0.44) | 0.07 (0.09)

ADVERSE EVENTS:
Time Frame: 2 sessions were held approximately 1 week apart. Adverse events were collected after receiving the first injection of study medication until 24 hours after the last session. This was approximately 8 days for participants assuming sessions were held one week apart.
Groups:
- Pain Group, Placebo Session: Patients with chronic pain who are maintained on methadone for opioid use disorder. Placebo: An IM injection of 0.9% normal saline will be given.
- Pain Group, Naloxone Session: Patients with chronic pain who are maintained on methadone for opioid use disorder. Naloxone Hydrochloride: An intramuscular (IM) injection of naloxone will be given.
- No Pain Group, Placebo Session: Patients who are maintained on methadone for opioid use disorder but who do not have chronic pain. Naloxone Hydrochloride: An intramuscular (IM) injection of naloxone will be given.
- No Pain Group, Naloxone Session: Patients who are maintained on methadone for opioid use disorder but who do not have chronic pain.
  Placebo: An IM injection of 0.9% normal saline will be given.
Arm/Group | Pain Group, Placebo Session | Pain Group, Naloxone Session | No Pain Group, Placebo Session | No Pain Group, Naloxone Session
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/6 | 2/6 | 1/4 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pain Group, Placebo Session (N=6) | Pain Group, Naloxone Session (N=6) | No Pain Group, Placebo Session (N=4) | No Pain Group, Naloxone Session (N=4)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tunnel Vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paranoia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye Irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
COVID-19 Public Health Emergency caused almost complete stoppage of research activities for over half of the grant time. We only had 10% of the proposed number of completers. Therefore, the decision was made to halt the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT04473950/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT04473950/ICF_001.pdf